CLINICAL TRIAL: NCT05157126
Title: A Masked, Randomized Controlled Trial Evaluating Locally-applied Gentamicin Versus Saline in Open Tibia Fractures
Brief Title: Gentamicin Open Tibia Study
Acronym: GO-Tibia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Muhimbili Orthopaedic Institute (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-35369; K23AR079044 (NIH)
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Fracture Open Tibia
MeSH Terms: interventions — Gentamicins; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single-center individually-randomized placebo-controlled superiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data collectors (research coordinators) and data analysts will also be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gentamicin (Experimental): The intervention consists of 80mg of liquid gentamicin diluted in 5 mL normal saline (16mg/mL). The solution is injected by inserting a 22-gauge needle down to bone through an anteromedial approach at the level of the fracture site such that the injected solution fills the wound cavity. A total of 5mL of study solution will be administered.
  Interventions: Drug: Gentamicin
- Saline (Placebo Comparator): The control consists of 5 mL normal saline injected immediately after wound closure at the open fracture site. The solution is injected by inserting a 22-gauge needle down to bone through an anteromedial approach at the level of the fracture site such that the injected solution fills the wound cavity. A total of 5mL of study solution will be administered.
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Gentamicin — Liquid gentamicin administered at the open fracture site
  Arms: Gentamicin
Drug: normal Saline — Normal saline administered at the open fracture site
  Arms: Saline

SUMMARY:
Local application of antibiotics directly to the traumatic wound is a promising treatment for the prevention of infection after open tibia fractures, which are a significant source of disease burden globally, particularly in low-income countries. This study aims to measure the effect of locally applied gentamicin on risk of infection for open tibial fractures in Tanzania. If proven effective, local gentamicin would be a highly cost-effective strategy to reduce complications and disability from open tibial fractures that could impact care in both high- and low-income countries.

DETAILED DESCRIPTION:
Tibial shaft (shinbone) fractures are the most common major fracture of the lower leg and are frequently associated with a break in the skin known as an open fracture. Because the bone is exposed by the open wound, open tibial fractures are often complicated by infection and failure of bone healing, which can lead to long-lasting disability and in some cases amputation. Intravenous antibiotics administered early after injury are a well-established measure to prevent fracture-related infection (FRI), but their effectiveness is limited by poor blood flow at the fracture site and inability to achieve high local concentrations with systemic administration. Gentamicin applied locally within the open fracture wound is a promising adjunctive measure to reduce the risk of FRI after these injuries, but there are no high-quality clinical trials evaluating its use.

This will be the first randomized trial evaluating locally administered gentamicin to reduce infection in a fracture population. If efficacious, local gentamicin is likely to be a highly cost-effective preventive strategy for FRI and may ultimately be cost saving. Although these findings will originate from a low-income country, results may be generalizable to populations in both high and low-income countries and could therefore significantly reduce the global burden of open fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Open tibial shaft fracture meeting the following criteria:

  1. Orthopaed Trauma Association (OTA) Type 42
  2. Primarily closable wound
  3. Gustilo-Anderson (GA) Type I, II, or IIIA

Exclusion Criteria:

* Time from injury to presentation > 48 hours
* Time from injury to surgery > 7 days
* Aminoglycoside allergy
* GA IIIB or IIIC open fractures
* Bilateral open tibial fractures
* Severe brain (GCS<12) or spinal cord injury
* Severe vascular injury
* Severe burns (>10% Total Body Surface Area (TBSA) or >5% TBSA with full thickness or circumferential injury)
* Pathologic fracture
* History of active limb infection, ipsilaterally
* Unlikely to complete follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of fracture-related infection (FRI) | 12 months
  Fracture-related infection is a consensus definition of infection after fracture treatment. It is diagnosed by an orthopaedic surgeon based on any of the following four diagnostic criteria: (1) fistula, sinus or wound breakdown; (2) purulent drainage from the wound or presence of pus during surgery; (3) phenotypically indistinguishable pathogens identified by culture from at least two separate deep tissue/implant specimens; or (4) presence of microorganisms in deep tissue taken during an operative intervention, as seen on histopathological examination.
  FRI diagnosis is likely to peak between 6 weeks and 6 months after surgery and has a non-normal time-to-event distribution, with incident cases rarely presenting later than 12 months after surgery. All events will be confirmed by an independent adjudication committee comprised of three masked, non-treating orthopaedic trauma surgeons.

SECONDARY OUTCOMES:
Occurrence of nonunion | 12 months
  Binary outcome based on the following criteria:
  1. Any unplanned reoperation for promotion of bone healing; OR
  2. Modified Radiographic Union Scale for Tibia Fractures (mRUST) ≤10 at 12 months follow-up AND either: Function IndeX for Trauma (FIX-IT) score ≤11 at 12 month follow-up, OR recommendation by treating surgeon for nonunion repair surgery
Occurrence of unplanned fracture-related reoperation | 12 months
  Occurrence of unplanned fracture-related reoperation, a binary variable, for infection, wound healing, or fracture union, excluding removal of implants for prominence/irritation. This may include but is not limited to:
  1. Irrigation and debridement of surgical incisions or open fracture wounds due to infections or wound healing problems;
  2. Revision wound closure for dehiscence;
  3. Soft tissue coverage procedure for infected or necrotic wound;
  4. Fracture delayed union or nonunion surgery (such as bone grafting or implant exchange);
  5. Reoperation for hardware or prosthesis failure due to infection or bone-healing problems;
  6. Amputation for infection, wound or fracture healing problem.
Health-related quality-of-life (HRQOL) as measured by EQ-5D-3L (Swahili version) | 12 months
  The EQ-5D is a survey instrument that assesses multiple domains of quality-of-life, including mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Fracture healing by modified Radiographic Union Scale for Tibial fractures (mRUST score) | 12 months
  The mRUST score is based on evaluation plain radiographs of the fracture site. Each cortex is scored from 1-4 based on the degree of healing and summed resulting in an ordinal scale ranging from 4 to 16, with higher score indicating greater fracture healing.
Clinical fracture healing by Function IndeX for Trauma (FIX-IT) | 12 months
  The FIX-IT score is an ordinal scale from 0-12 that encompasses two domains: ability to weight-bear and pain at fracture site, each scored from 0-6. Higher score indicates more clinical healing.
Occurence of FRI Suggestive Criteria | 12 months
  Suggestive criteria are signs/symptoms of infection that do not meet criteria for definitive fracture-related infection (FRI). These include clinical signs (wound redness, fever) and radiographic signs (sequestrum), elevated serum inflammatory markers, and new onset or increased non-purulent wound drainage.

OTHER OUTCOMES:
Adverse events | 12 months
  All serious and non-serious adverse events will be reported as counts for each treatment group
Fold-change in creatinine level | 2 days
  Creatinine is a laboratory value used to assess kidney function. Creatinine levels will be measured preoperatively and 2-days postoperatively for all study participants.

CONTACTS AND LOCATIONS:
Overall Officials: David W Shearer, MD, MPH, Principal Investigator — University of California, San Francisco; Billy T Haonga, MD, Principal Investigator — Muhimbili Orthopaedic Institute
Locations (1):
- Muhimbili Orthopaedic Institute, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haonga BT, O'Marr JM, Ngunyale P, Ngahyoma J, Kessey J, Sasillo I, Rodarte P, Belaye T, Berhaneselase E, Eliezer E, Porco TC, Morshed S, Shearer DW. GO-Tibia: a masked, randomized control trial evaluating gentamicin versus saline in open tibia fractures. Trials. 2023 Jun 15;24(1):406. doi: 10.1186/s13063-023-07410-0. PMID 37322521